CLINICAL TRIAL: NCT06702345
Title: Establishing a Clostridioides Difficile Controlled Human Infection Model
Brief Title: Clostridioides Difficile Controlled Human Infection Model
Acronym: CloDiCHI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Helmholtz Centre for Infection Research (Other); GlaxoSmithKline (Industry); University of Oxford (Other); University of Cologne (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof. dr. M. Roestenberg, Leiden University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CloDiCHI; Grant number: 101007799 (Other Grant/Funding Number: Innovative Health Initiative)
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: C. Difficile; C. Difficile Infection; Controlled Human Infection
MeSH Terms: interventions — Vancomycin; Clindamycin

STUDY DESIGN:
Intervention Model Description: This will be a first in human, open-label, adaptive design, escalating clinical trial, investigating the oral exposure of toxigenic C. difficile in healthy volunteers. The adaptive design is aimed at a stepwise escalation to ensure safety of trial participants and gear towards the optimal balance between endpoints and tolerability. The study will start with one cohort of volunteers, cohort A, with an option to escalate to a second cohort, cohort B, and a third cohort, cohort C, if needed. Escalation to the subsequent cohort will be performed by adding antibiotic pretreatment. Escalation will be based upon safety first and secondly upon microbiological and clinical endpoints (ideally aiming for an attack rate of 70% in both). In every cohort small pilot groups (of five volunteers each) will be used to flag safety signals and determine the escalation schedule, having the option to include 15 more participants to the same cohort or escalate to the pilot group of the subsequent cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (TCD spores only) (Experimental): Volunteers in cohort A will be exposed to a once a day capsule with 10^4 CFU TCD spores for 12 days. First, a pilot group of 5 volunteers will be exposed to flag safety signals. If in this pilot group TCD exposure is well tolerated and less than 70% of the volunteers (< 4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, the trial will escalate to the second cohort, cohort B. If, however, in the pilot group TCD exposure is well tolerated and at least 70% of the volunteers (≥4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, a confirmatory group of another 15 volunteers will be included in cohort A (total 20 volunteers). If in this total of 20 volunteers sat least 70% (≥ 14 out of 20 volunteers) reaches a clinical AND microbiological endpoint, no further escalation to cohort B or C will be done. If, however, less than 70% of the 20 volunteers in cohort A reaches a clinical AND microbiological endpoint, escalation will continue to cohort B.
  Interventions: Other: encapsulated 10^4 CFU toxigenic. C. difficile spores
- Cohort B (vancomycin pretreatment + TCD spores) (Experimental): Volunteers in cohort B will be exposed first to 5 days of oral vancomycin pretreatment, 4 times a day 250mg, followed immediately by once a day capsule with 10^4 CFU TCD spores for 12 days. First, a pilot group of 5 volunteers will be exposed to flag safety signals. If in this pilot group TCD exposure is well tolerated and less than 70% of the volunteers (< 4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, the trial will escalate to the third cohort, cohort C. If, however, in the pilot group TCD exposure is well tolerated and at least 70% of the volunteers (≥4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, a confirmatory group of another 15 volunteers will be included in cohort B (total 20 volunteers). If in this total of 20 volunteers at least 70% (≥ 14 out of 20 volunteers) reaches a clinical AND microbiological endpoint, no further escalation to cohort C will be done. If, however, this is less then 70%, escalation continues to cohort C.
  Interventions: Other: encapsulated 10^4 CFU toxigenic. C. difficile spores; Drug: Vancomycin
- Cohort C (clindamycin pretreatment + TCD spores) (Experimental): Volunteers in cohort C will be exposed first to five days of oral clindamycin pretreatment, three times a day 600mg, followed immediately by once-a-day dosing of 104 CFU TCD spores (capsules) for 12 consecutive days. First, a small pilot group of five volunteers will be exposed to flag safety signals. If in this pilot group TCD exposure is well tolerated and less than 70% of the volunteers (< 4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, the trial will stop. If, however, in the pilot group TCD exposure is well tolerated and at least 70% of the volunteers (≥4 out of 5 volunteers) reaches a microbiological AND clinical endpoint, a confirmatory group of another 15 volunteers will be included in cohort C (total 20 volunteers), after which the trial will stop.
  Interventions: Other: encapsulated 10^4 CFU toxigenic. C. difficile spores; Drug: Clindamycin

INTERVENTIONS:
Other: encapsulated 10^4 CFU toxigenic. C. difficile spores — 12 consecutive days of once a day a capsule with 10^4 CFU toxigenic C. difficile spores.
Drug: Vancomycin — oral vancomycin pretreatment, 4 times a day 250mg, given the five days before toxigenic C. difficile exposure.
  Arms: Cohort B (vancomycin pretreatment + TCD spores)
Drug: Clindamycin — oral clindamycin pretreatment, 3 times a day 600mg, given the five days before toxigenic C. difficile exposure
  Arms: Cohort C (clindamycin pretreatment + TCD spores)

SUMMARY:
This study will investigate in healthy study subjects, the safety and tolerability of a controlled infection with Clostridioides difficile, a gut bacterium that can cause diarrhoea. It is also examined which dosing regimen (with or without antibiotic pretreatment) is required to induce mild symptoms (like diarrhoea) in the majority of study subjects and which microbiota and immunological factors influence this.

To investigate this, healthy adult study subjects will be asked to ingest capsules (pills) containing the Clostridioides bacterium.

DETAILED DESCRIPTION:
This will be a first in human, open-label, adaptive clinical trial investigating the oral exposure of toxigenic C. difficile in healthy volunteers. The trial will consist of at least one cohort (cohort A), with an option to escalate to a second (cohort B) and third cohort (cohort C) if needed. In every cohort volunteers will be exposed for 12 consecutive days (D0-D11) to once a day a capsule with 10^4 CFU toxigenic C. difficile spores. Escalation will be done by adding antibiotic pretreatment (vancomycin in cohort B and clindamycin in cohort C) the five days before C. difficile exposure (D-6 - D-1). Escalation will be based upon safety first and secondly upon microbiological and clinical endpoints (ideally aiming for a 70% attack rate in both). In every cohort there will be first a pilot group of 5 volunteers, after which there is an option to include a confirmatory group of 15 more participants in the same cohort if the exposure is safe and the threshold for the microbiological and clinical endpoint is met.

Immediately following the first ingestion of the C. difficile spores (day 0), volunteers will be closely and strictly monitored for adverse events (AEs) and vital signs in an outpatient setting. Until day 35, AEs, vital signs and stool samples for C. difficile toxin PCR/EIA, culture, and microbiota analysis will be collected every other day, safety laboratory measurements will be performed once in four days (starting from day 0). Immunology samples will be collected on day 0, 2, 20, 35 and 84. If a volunteer develops symptoms of CDI the volunteer needs to visit the research clinic the same day for a physical check-up, and collection of a blood and stool sample, and, if needed (antibiotic) treatment will be started according to standard of care. Any recurrent episode of a C. difficile infection will be treated with fecal microbiota transplantation (FMT). A final visit will take place after three months (day 84), with collection of feces and blood. If a volunteer is still C. difficile positive at this timepoint, they will be followed every three months until decolonisation is reached, up to a maximum of one year after the start of the trial. Decolonisation will be de-fined as having a negative molecular C. difficile test on at least two different timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥18 and ≤45 years and in good health;
2. Body mass index (BMI) ≥18.0 and <30.0 kg/m2;
3. Subject has adequate understanding of the procedures of the study and is able and willing to abide strictly thereby;
4. Subject is able to communicate well with the investigator, is willing to follow hygienic measures and instructions;
5. For women of childbearing potential: subject agrees to use adequate contra-ception (see Appendix D for the different adequate contraception methods for this study) and not to breastfeed for the duration of the study;
6. Subject has signed informed consent.

Exclusion Criteria:

1. Any physical or psychiatric illness or conditions that could threaten or com-promise the health of the subject during the study, influence their ability to par-ticipate in the trial or interfere with the interpretation of the study results, as de-termined by the trial physician;
2. Use of systemic (IV or oral) antibiotics within three months prior to screening; other microbiota influencing medication (that could influence the trial, based on the Investigator's opinion) within 1 month prior to screening visit. Prior use of topical antibiotics is permitted if there is no clinically relevant systemic ex-pected following assessment of the trial physician and are expected to be dis-continued during the start of the first study activity.
3. Has had a recent hospitalization (e.g. 3 months prior to screening) and/or has someone in immediate social circle who is frequently hospitalized (≥3 times in a 12-month period) or frequently exposed to hospital settings (≥ one time a month, e.g. dialysis units);
4. Regular use (defined by more than once weekly) of proton-pump inhibitors or H2-blockers during one month prior to screening;
5. Chronic use of immunosuppressive drugs, e.g. systemic corticosteroids or other immune modifying drugs (with exception of oral anti-histamines and top-ical/inhaled corticosteroids);
6. Positive HIV, Hepatitis B or C screening tests;
7. Known immunodeficiency disorders;
8. The use of strong P-glycoprotein-inhibitors (like ciclosporin, ketoconazole, erythromycin, clarithromycin, verapamil and amiodaron) during the trial;
9. Known allergy to vancomycin, clindamycin, fidaxomicin (and macrolides), or metronidazole;
10. Any known significant allergy against the excipients of C. difficile inoculum or inability to swallow capsules;
11. Known gastro-intestinal disease including but not limited to inflammatory bow-el diseases (Crohn's disease, Colitis ulcerosa), a history of bowel resection or any other gastro-intestinal surgery which has significantly changed the ana-tomical structure or physiological function of the gastro-intestinal tract, bile ac-id secretion abnormalities, constipation defined by bowel movements less than every second day or chronic use of laxatives;
12. Positive fecal culture or PCR with toxigenic or non-toxigenic Clostridioides spp. or SSYC (Salmonella spp., Shigella spp., Yersinia spp. or Campylobac-ter spp.) at screening, or recent (<14 days) history of diarrhoea (i.e. as ≥3 loose stools (Bristol stool scale 6-7) in 24 hours);
13. Any condition that would put household members or close contacts at a great-er risk for transmission e.g. no access or use of flush toilet;
14. Individuals living, working or having close contact with people who belong to vulnerable populations such as hospitalized patients, pregnant women, im-mune compromised individuals, children younger than 2 years, residents of nursing homes, elderly older than 70 years of age, or any person with a medi-cal condition at risk of developing severe CDI.
15. Individuals working in food preparation;
16. Individuals having close contact with healthcare personal/individuals working in food preparation;
17. For women of childbearing potential; a positive serological pregnancy test at screening or lactating at screening/ during the trial;
18. History of drug or alcohol abuse interfering with normal social functioning in the period of one year prior to study onset, positive urine toxicology test for il-licit drug use at screening;
19. Receipt of another investigational agent within 90 days prior or 60 days after C. difficile ingestion;
20. Any condition or situation that could influence the independent consent of par-ticipant (e.g. being a direct colleague or family member of study personnel).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of exposure to toxigenic C. difficile spores with optional antibiotic pretreatment | from day 0 until day 35 for cohort A and from day -5 until day 35 for cohort B and C.
  number and grade of (related) adverse events
Colonisation with the challenge C. difficile strain | on at least two timepoints from day 14 until day 35
  1. Proven: a positive culture of toxigenic C. difficile with the same molecular identity as the challenge strain, without symptoms of CDI.
  2. Probable: a positive toxin EIA on stool samples OR a positive feces tcdB-PCR, without symptoms of CDI.
Infection with the challenge C. difficile strain | from day 0 until day 35
  1. Proven: clinical findings compatible with CDI (clinical findings should include at least diarrhoea: Bristol stool chart type 6-7 plus ≥ 3 stools in 24 hours) and a positive culture of toxigenic C. difficile with the same molecular identity as the challenge strain
  2. Probable: clinical findings compatible with CDI (clinical findings should include at least diarrhoea: Bristol stool chart type 6-7 plus ≥ 3 stools in 24 hours) and a positive toxin EIA on stool samples OR a positive feces tcdB-PCR

SECONDARY OUTCOMES:
Colonisation with a non-challenge C. difficile strain | on at least two timepoints from day 14 until day 35
  Proven microbiological endpoint/colonisation with non-challenge strain: a positive culture of C. difficile with another molecular identity than the challenge strain, without symptoms of CDI.
Infection with non-challenge C. difficile strain | from day 0 until day 35
  Clinical findings compatible with CDI (clinical findings should include at least diarrhoea: Bristol stool chart type 6-7 plus ≥ 3 stools in 24 hours) and a positive culture of C. difficile with another molecular identity than the challenge strain
Kinetics of C. difficile colonisation/infection over time | from day 0 until day 35
  Quantitative measurement of C. difficile by qPCR at samples taken every other day
Systemic immune response following C. difficile colonisation and/or infection | at day 0, 20, 35 and 84.
  Anti-Toxin A and anti-Toxin B neutralizing antibody titers by toxin neutralization assay (TNA) on serum samples
Antibody response following C. difficile colonisation and/or infection | at day 0, 20, 35, 84 and first day of C. difficile infection symptoms.
  ELISA for antibody responses against various antigens in serum and faecal samples
Cytokine response related to C. difficile colonisation and/or infection | at day 0, 2, 20 and first day of C. difficile infection symptoms.
  Cytokine measurement in serum and faecal samples
Calprotectin and potential other biomarkers related to C. difficile colonisation and/or infection | on day 0, 20 and 35
  Calprotectin and potential other biomarkers for inflammation (like lactoferrin) in faecal samples

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No